CLINICAL TRIAL: NCT00024921
Title: The Genetics of Kidneys in Diabetes (GoKinD) Study
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Other Study IDs: NCRR-M01RR00036-0805
Record Dates: First submitted 2001-10-05; First posted 2001-10-10 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2003-12

CONDITIONS: Diabetic Nephropathy
MeSH Terms: conditions — Diabetic Nephropathies

SUMMARY:
Kidney disease in diabetes (diabetic nephropathy) tends to run in families. It is likely, therefore, that there are genes that predict or are associated with either getting or not getting diabetic nephropathy. The GoKinD Study will provide clinical information and DNA for investigators to look for these genes. Evaluation will be performed and DNA obtained from approximately 1100 diabetic persons with kidney disease and 1000 diabetic persons without kidney disease. In some cases, samples for DNA will also be obtained from the parents of these subjects. Clinical information and DNA will be coded so that individuals cannot be identified, but the DNA can be linked to the clinical data from the individual. Multiple investigators will be able to use this genetic material to test hypotheses about the genetics of kidney disease in diabetes.

ELIGIBILITY:
Inclusion criteria:

Type 1 diabetes mellitus with or without diabetic nephropathy; 19-54 years old; no other kidney disease

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2100 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University, St Louis, Missouri, United States